CLINICAL TRIAL: NCT04234152
Title: Complete Shielding of Multivitamins to Reduce Toxic Peroxides in the Parenteral Nutrition: A Pilot Study (C SMART-PN, Pilot)
Brief Title: Complete Shielding of Multivitamins to Reduce Toxic Peroxides in the Parenteral Nutrition: A Pilot Study
Acronym: C-SMART-PN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Ibrahim Mohamed, Paediatrician-Neonatologist, Associate professor of Paediatrics and Nutrition, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-2713
Record Dates: First submitted 2020-01-08; First posted 2020-01-21 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Parenteral Nutrition; Infant, Premature, Diseases; Infant, Newborn, Disease; Lung Diseases; Respiratory Tract Disease; Bronchopulmonary Dysplasia; Pathologic Processes
Keywords: Photo-protection of Multivitamins; Oxidative Stress; Ascorbyl peroxide; Urine peroxides
MeSH Terms: conditions — Hyperphagia; Infant, Premature, Diseases; Disease; Lung Diseases; Respiratory Tract Diseases; Bronchopulmonary Dysplasia; Pathologic Processes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome is the concentration of peroxides in the urine. The urine samples will not indicate the arm of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MV Photo-protection (Experimental): Includes infants in whom the new procedure of MV separation and photo-protection will be applied. This arm will be stratified to male and female 1:1
  Interventions: Other: Photo-protection
- Standard of care (Placebo Comparator): Includes infants in whom the standard method of preparation and infusion of PN will be applied. This arm will be stratified to male and female 1:1
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Photo-protection — The MV solution is delivered from producing companies in amber vials. The MV will be sampled by the pharmacy technician in a syringe that is photo-protected with a white label indicating the subject study name, protocol number and the infusion rate. The MV will be transported to the unit in the same photo-protected syringe. In the neonatal unit, this syringe will be installed in the pump and connected to photo-protected extension duration.
  Arms: MV Photo-protection
Other: Standard Care — This group will receive the standard practice of PN compounding in the pharmacy followed by infusion in standard infusion kit available in Sainte-Justine's Hospital.
  Arms: Standard of care

SUMMARY:
The purpose of this study is to examine if a new and simple method involving complete photo-protection of multivitamins only (since sampling through infusion) will result in a significant reduction of peroxide contamination of parenteral nutrition compared to standard method of parenteral nutrition preparation and infusion in extremely preterm infants.

DETAILED DESCRIPTION:
Hypothesis and Objectives:

The investigators propose, in this pilot study, a new and simple method involving complete photo-protection of multivitamins (MV) only (since sampling through infusion) and they hypothesize that this method will be readily applicable and will result in a significant reduction of peroxide contamination of parenteral nutrition (PN) compared to standard care of PN preparation and infusion method.

In Vitro Results Using This Proposed Photo-Protection Method:

This method has reduced the quantity of infused peroxides (as equivalent H2O2). When adding the generated peroxides over 5 hours (5 samples: at times 0, 30 minutes, 1, 3 and 5 hours), the total peroxides were 1270± 47 micromolar (μM) without photo-protection vs. 710±16 μM with this method, leading to 45% reduction of peroxides (data presented as a poster presentation in the Pediatric academic societies meeting , 2018, Poster number 2874.625). This reduction is comparable to the previously reported in vitro data for the whole PN complete photo-protection that reported 50% reduction of peroxides.

Specific objective of this pilot study:

To examine if this new and simple method will be feasible in clinical practice and will result in a significant reduction of urinary peroxide concentration when compared to standard PN compounding and infusion technique.

Innovation:

The investigators' team's long experience in this field permitted the identification of the interaction between light and MV (specifically riboflavin) that leads to doubling the amount of peroxides contaminating the PN. The complexity of complete photo-protection encountered by the team to conduct small uni-center studies and the incapacity to introduce the complete photo-protection in daily clinical practice led the team to create this simple intervention that will address the problem at its origin in a practical way. All trials, including complete PN photo-protection, faced the complexity of keeping MV away from light while needing to prepare the PN admixture under the light of a sterile hood. Added to this was the complexity of completely covering the PN bag while compounding the admixture. Light exposure may also occur during the transportation of the PN from the hospital pharmacy to the neonatal unit (even with special attention to the bottom of the bag and the area around the tubing being well covered).

The proposed intervention will eliminate all these complex procedures by directly sampling the MV in a photo-protected syringe, transporting it in this syringe, and directly infusing the MV into the photo-protected intravenous lines through its infusion into the patient.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 28 weeks of gestational age
* Obtaining parental consent before the start of the first PN prescribed by the attending physician

Exclusion Criteria:

* Significant congenital malformations
* Infant is currently enrolled in another trial -unless approval of trial research team-
* Parent inability to comprehend and consent

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Change in urine peroxides concentration | Baseline, 48 hours post-parenteral nutrition and on day 7 of life
  From each urine sample, an aliquot (0.2 ml) will be used for creatinin measurement whereas another (0.5 ml) will be used for peroxide determination using the ferrous oxidation/xylenol orange technique. H2O2 will serve for the standard curve. The results will be expressed as μmol equ H2O2/mg creatinine.

SECONDARY OUTCOMES:
Urinary ascorbylperoxide (AscOOH) | On day 7 of life
  Urine AscOOH concentration will be determined using Mass spectrometry.
Whole blood glutathione redox potential | On day 7 of life
  Whole blood levels of glutathione (GSH) and glutathione disulfide (GSSG) will be measured by capillary electrophoresis as previously described by the investigators' team, using 0.5 ml of blood. The whole blood redox potential (mV) will be calculated, using the Nernst equation.
Whole blood glutathione redox potential | At 36 weeks Post-Menstrual Age
  Whole blood levels of glutathione (GSH) and glutathione disulfide (GSSG) will be measured by capillary electrophoresis as previously described by our team, using 0.5 ml of blood. The whole blood redox potential (mV) will be calculated, using the Nernst equation.
Serum inflammatory cytokines: Interleukin 1 alpha (IL-1alpha) and beta (IL-1beta), Interleukin 6 (IL-6), Interleukin 8 (IL-8), Interleukin (IL-10), Tumor Necrosis Factor alpha (TNF-alpha), Vascular Endothelial Growth Factor (VEGF) | On day 7 of life
  Multiplex assay (Luminex R&D systems), using 0.1 ml of blood
Serum inflammatory cytokines: IL-1alpha, IL-1beta, IL-6, IL-8, IL-10, TNF-alpha, VEGF | At 36 weeks Post-Menstrual Age
  Multiplex assay (Luminex R&D systems), using 0.1 ml of blood
Clinical outcome - Incidence of Bronchopulmonary dysplasia (BPD) and BPD severity (Mild, moderate, sever) | At 36 weeks Post-Menstrual Age
  According to the National Institute of Child Health and Human Development (NICHD) criteria (Jobe Alan H.,2001)
Clinical outcome - Mortality rate | At 36 weeks Post-Menstrual Age
  Death before 36 weeks post menstrual age
Clinical outcome - length of mechanical ventilation (invasive, non-invasive) | From birth to discharge home, an average of 4 months
  Total number of days on mechanical ventilation (both invasive and non invasive respiratory support)
Clinical outcome - length of supplemental oxygen (in days) | From birth to discharge home, an average of 4 months
  Total number of days on Nasal cannula O2 supplements
Clinical outcome - Incidence and stage of necrotizing enterocolitis (According to Bell's classification) | From birth to discharge home, an average of 4 months
  Necrotizing enterocolitis stages as defind by Bell stage II or higher. The incidence in the two arms will be reported and compared
Clinical outcome - Incidence and grade of intraventricular hemorrhage (IVH), according to Papille criteria | From birth to discharge home, an average of 4 months
  Any intraventricular hemorrhage (IVH), IVH grade III and IV in each arm will be reported and compared.
Clinical outcome - Incidence of significant liver cholestasis (defined as two or more consecutive conjugated bilirubin values ≥ 34 μmol/L) | From birth to discharge home, an average of 4 months
  Cholestasis is defined as two or more consecutive conjugated bilirubin values ≥ 34 μmol/L. The incidence of cholestasis in each arm will be reported and compared.
Clinical outcome - Incidence and stage of Retinopathy Of Prematurity (ROP) (highest stage) | From birth to discharge home, an average of 4 months
  The incidence of ROP stage II and higher as defined by the National Eye Institute will be reported and compared.
Clinical outcome - Incidence of significant Patent Ductus Arteriosus (PDA) | From birth to discharge home, an average of 4 months
  PDA requiring medical or surgical treatment according to the treating neonatologist will be reported and compared.
Clinical outcome - infant anthropometry: weight | At 36 weeks Post-Menstrual Age
  Weight in grams
Clinical outcome - infant anthropometry: length | At 36 weeks Post-Menstrual Age
  Length in centimeters
Clinical outcome - infant anthropometry: head circumference | At 36 weeks Post-Menstrual Age
  Head circumference in centimeters
Clinical outcome - length of hospital stay (in days) | From birth to discharge home, an average of 4 months
  Total number of days till discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Mohamed, M.D.,Ph.D., Principal Investigator — Sainte-Justine Research center, Sainte-Justine hospital, University of Montreal
Locations (2):
- Canada (2):
  - CHU Sainte-Justine, Montreal, Quebec
  - University of Montreal, Sainte-Justine Hospital, Montreal

IPD SHARING:
Plan to Share IPD: Yes
The authors will do every efforts to make the study protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR) and analytic code available to other researcher (either by protocol publication before the study of as supplemental material with the final publication).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of collecting all data and for a maximum of 2 years
Access Criteria: Anonymized information will be available for research and academic purposes.

REFERENCES:
- [Background] Thibeault DW. The precarious antioxidant defenses of the preterm infant. Am J Perinatol. 2000;17(4):167-81. doi: 10.1055/s-2000-9422. PMID 11041438
- [Background] Mohamed I, Elremaly W, Rouleau T, Lavoie JC. Oxygen and parenteral nutrition two main oxidants for extremely preterm infants: 'It all adds up'. J Neonatal Perinatal Med. 2015;8(3):189-97. doi: 10.3233/NPM-15814091. PMID 26485550
- [Background] Saugstad OD. Oxygen and oxidative stress in bronchopulmonary dysplasia. J Perinat Med. 2010 Nov;38(6):571-7. doi: 10.1515/jpm.2010.108. Epub 2010 Aug 31. PMID 20807008
- [Background] Laborie S, Lavoie JC, Pineault M, Chessex P. Contribution of multivitamins, air, and light in the generation of peroxides in adult and neonatal parenteral nutrition solutions. Ann Pharmacother. 2000 Apr;34(4):440-5. doi: 10.1345/aph.19182. PMID 10772427
- [Background] Laborie S, Lavoie JC, Chessex P. Increased urinary peroxides in newborn infants receiving parenteral nutrition exposed to light. J Pediatr. 2000 May;136(5):628-32. doi: 10.1067/mpd.2000.105131. PMID 10802495
- [Background] Bassiouny MR, Almarsafawy H, Abdel-Hady H, Nasef N, Hammad TA, Aly H. A randomized controlled trial on parenteral nutrition, oxidative stress, and chronic lung diseases in preterm infants. J Pediatr Gastroenterol Nutr. 2009 Mar;48(3):363-9. doi: 10.1097/mpg.0b013e31818c8623. PMID 19274793
- [Background] Mohamed I, Elremaly W, Rouleau T, Lavoie JC. Ascorbylperoxide Contaminating Parenteral Nutrition Is Associated With Bronchopulmonary Dysplasia or Death in Extremely Preterm Infants. JPEN J Parenter Enteral Nutr. 2017 Aug;41(6):1023-1029. doi: 10.1177/0148607116643704. Epub 2016 Apr 1. PMID 27036126
- [Background] Elremaly W, Mohamed I, Mialet-Marty T, Rouleau T, Lavoie JC. Ascorbylperoxide from parenteral nutrition induces an increase of redox potential of glutathione and loss of alveoli in newborn guinea pig lungs. Redox Biol. 2014 May 20;2:725-31. doi: 10.1016/j.redox.2014.05.002. eCollection 2014. PMID 25009773
- [Background] Lavoie JC, Rouleau T, Chessex P. Interaction between ascorbate and light-exposed riboflavin induces lung remodeling. J Pharmacol Exp Ther. 2004 Nov;311(2):634-9. doi: 10.1124/jpet.104.070755. Epub 2004 Jul 13. PMID 15254143
- [Background] Chessex P, Harrison A, Khashu M, Lavoie JC. In preterm neonates, is the risk of developing bronchopulmonary dysplasia influenced by the failure to protect total parenteral nutrition from exposure to ambient light? J Pediatr. 2007 Aug;151(2):213-4. doi: 10.1016/j.jpeds.2007.04.029. PMID 17643781
- [Background] Chessex P, Laborie S, Nasef N, Masse B, Lavoie JC. Shielding Parenteral Nutrition From Light Improves Survival Rate in Premature Infants. JPEN J Parenter Enteral Nutr. 2017 Mar;41(3):378-383. doi: 10.1177/0148607115606407. Epub 2016 Sep 30. PMID 26376662